CLINICAL TRIAL: NCT03183856
Title: Comparison of Clinical Efficacy and Safety for Ambulatory and Functional Improvement in Patients After Total Knee Arthroplasty With Morning Walk
Brief Title: Comparison of Ambulatory and Functional Improvement by Morning Walk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulsan University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Chang Ho Hwang, PhD and MD, Ulsan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: chhwang7
Record Dates: First submitted 2017-06-06; First posted 2017-06-12 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Arthroplasty, Replacement, Knee; Robotics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning walk (Experimental): 200 steps of gait rehabilitation using an end-effector typed gait robot with 5 minute break, 3 times a day for 10 weekdays: the end-effector type gait robot (Morning Walk®, Hyundai Heavy Industry, Republic of Korea)
  Interventions: Device: Morning walk
- No Morning walk (Active Comparator): 200 steps by themselves or with a help of a walker on a even floor at a comfortable pace with 5 minute break, three times a day for 10 weekdays
  Interventions: Other: no Morning walk

INTERVENTIONS:
Device: Morning walk — a end-effector typed gait robot with a saddle
  Arms: Morning walk
Other: no Morning walk — ambulation voluntary or with a help of walker
  Arms: No Morning walk

SUMMARY:
The aim of this study is to determine the clinical efficacy and feasability of gait rehabilitation robot through approving functional improvement by an end-effector typed gait robot in patients underwent total knee arthroplasty.

DETAILED DESCRIPTION:
pre-interventional evaluation; within 1 day of initiation of the intervention; 5 days after initiation of the intervention; 10 days after intervention after initiation of the intervention; 42 days after intervention start

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent Unilateral or both Total Knee Arthroplasty

Exclusion Criteria:

* brain disease, spinal cord injury, peripheral neuropathy, myopathy
* Inability to ambulate fully due to muscukoskeletal disorders
* MMSE<23
* history of arthroplasty surgery on either of legs
* Cardiac pacemaker
* Refusal of participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Change of WOMAC index | 1 day before the initiation of intervention), 5 day, 10 day, and 31 days after the initiation of intervention
  Western Ontario and McMaster Universities Osteoarthritis Index

SECONDARY OUTCOMES:
Change of VAS | 1 day before the initiation of intervention), 5 day, 10 day, and 31 days after the initiation of intervention
  visual analogue scale

OTHER OUTCOMES:
Change of ROM | 1 day before the initiation of intervention), 5 day, 10 day, and 31 days after the initiation of intervention
  range of motion of the operated knee
Change of drug consumption | 5 day, and 10 day after the initiation of intervention
  weekly amount of tridol consumption
Change of 6 minute walk test | 1 day before the initiation of intervention), 5 day, 10 day, and 31 days after the initiation of intervention
  6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D., Ph.D., Study Director — Ulsan University Hospital
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea

IPD SHARING:
Plan to Share IPD: No